CLINICAL TRIAL: NCT02645461
Title: Acetylcholine Receptors From Human Muscles as Pharmacological Target for ALS
Acronym: AchALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Maurizio Inghilleri, Associated Professor of Neurology, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 3314
Record Dates: First submitted 2015-12-22; First posted 2016-01-01 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Riluzole (Active Comparator): Riluzole 50 mg twice daily in ALS patients
  Interventions: Drug: Riluzole
- PEA plus Riluzole (Experimental): Riluzole 50 mg twice daily plus Endocannabinoid palmitoylethanolamide (PEA) (ultramicronized) 600 mg twice daily in ALS patients
  Interventions: Drug: endocannabinoid palmitoylethanolamide (PEA); Drug: Riluzole

INTERVENTIONS:
Drug: endocannabinoid palmitoylethanolamide (PEA) — Endocannabinoid palmitoylethanolamide (PEA) (ultramicronized) 600 mg twice daily
  Other Names: PEA
  Arms: PEA plus Riluzole
Drug: Riluzole — Riluzole 50 mg twice daily

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a fatal disease leading to motor neuron degeneration and progressive paralysis. Other studies have revealed defects in skeletal muscle even in absence of motor neuron anomalies, focusing on acetylcholine receptors (AChRs) and supporting the so-called "dying-back" hypothesis. Outcome of this study will be to understand if the endocannabinoid palmitoylethanolamide (PEA) can reduce the rundown of AChRs currents in ALS muscle, and if it can modify ALS patients' clinical and electrophysiological parameters.

DETAILED DESCRIPTION:
Outcome:

Monitoring the efficacy and safety of PEA in the treatment of patients with ALS. Analysis of AChR currents and description of the composition of AChRs subunits in ALS muscles

Design of the Study:

A randomized controlled blinded study. Patients with sporadic ALS will receive riluzole alone or riluzole+PEA in order to investigate the clinical and electrophysiological effects of treatment. The expected number of enrolled patients will be 50.

All patients satisfying the selection criteria will be randomized into two groups: a first group will be treated only with riluzole, the second group with riluzole associated with PEA (Normast 600 mg microgranular, 2 sachets/day). The randomization will be done stratifying patietns according to type of clinical onset (bulbar vs. spinal). The patients will be enrolled in the Department of Neurology and Psychiatry, University of Rome "Sapienza".

The visits will be performed at 0 (randomization), 3 and 6 months. At each visit the ALS Functional Rating Scale-Revised (ALSFRS-R), the percentage of predicted forced vital capacity (FVC%), the Medical Research Council (MRC) score for muscle strength limited to the right upper limbs, and the compound muscle action potentials (CMAP) from right ulnar and phrenic nerves will be assessed. A muscle biopsy will be done at the end of the study. The obtained results will be compared with those observed in muscle samples from denervated (non-ALS) control patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALS according to the El-Escorial criteria;
* Age> 18 years;
* ALS Functional Rating Scale-Revised (ALSFRS- r) score> 20;
* Forced Vital Capacity (FVC)> 30%;
* Treatment with Riluzole.

Exclusion Criteria:

* Other diseases motor neurons;
* Experimental treatments in the previous three months;
* Pregnant or breast-feeding;
* Contraindications to the use of riluzole;
* Patients undergoing tracheostomy, enteral or parenteral supply;
* Severe psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in pulmonary capacity of ALS patients at 6 months. | six months
  Changes of the percentage of predicted forced vital capacity (FVC %) will be measured

SECONDARY OUTCOMES:
Changes in acetylcholine receptors (AChR) currents and Analysis of the composition of AChRs subunits in ALS muscles. | six months
  Utilization of voltage-clamp intracellular recordings in oocytes transplanted with membranes from ALS muscles.
Changes from baseline in muscle strength of ALS patients at 6 months. | six months
  Changes of the Medical Research Council (MRC) scale score will be measured
Changes from baseline in electrophysiological parameters of ALS patients at 6 months | six months
  Changes of the compound muscle action potential (CMAP) amplitude of ulnar and phrenic nerves will be measured